CLINICAL TRIAL: NCT05569304
Title: Endoscopic Sleeve Gastroplasty Versus GLP-1 Analogue for Class 1 and 2 Obesity Study (EGG Study)
Brief Title: Endoscopic Sleeve Gastroplasty Versus GLP-1 Analogue for Class 1 and 2 Obesity Study
Acronym: EGG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sengkang General Hospital (Other)
Responsible Party: Principal Investigator, Chue Koy Min, Associate Consultant, Sengkang General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIRB Ref: 2022/2469
Record Dates: First submitted 2022-10-04; First posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic Sleeve Gastroplasty Arm (Experimental): Prospective cohort of patients with classes 1 and 2 obesity that had consented to undergo endoscopic sleeve gastroplasty.
  Interventions: Procedure: Endoscopic sleeve gastroplasty
- Retrospective cohort (No Intervention): Retrospective cohort of patients with classes 1 and 2 obesity who did not undergo endoscopic sleeve gastroplasty and had been put on GLP-1 analogues

INTERVENTIONS:
Procedure: Endoscopic sleeve gastroplasty — Endoscopic sleeve gastroplasty
  Arms: Endoscopic Sleeve Gastroplasty Arm

SUMMARY:
The aim of this study is to compare the 1-year total body weight loss outcomes for Class 1 and Class 2 Obesity patients who have undergone endoscopic sleeve gastroplasty (ESG) in contrast to medical treatment with glucagon-like peptide-1 (GLP-1) analogues.

DETAILED DESCRIPTION:
Endoscopic sleeve gastroplasty (ESG) was developed with the aim of emulating the successful outcomes observed with sleeve gastrectomy, while obviating the need to permanently remove a large portion of the stomach. The recent MERIT trial reported that the estimated total body weight loss after ESG at 1-year was 13.6%, demonstrating superiority over lifestyle modifications alone.

Glucagon-like peptide-1 (GLP-1) analogues such as liraglutide or semaglutide are currently approved for the treatment of obesity and type 2 diabetes mellitus. Evidence supports the use of these medications in weight loss. The total body weight loss from GLP-1 analogues reportedly range between 7.8-13.8%.

As such, for patients with type 1 or 2 obesity who may not be candidates for bariatric surgery, the reported total body weight loss attainable by ESG and GLP-1 analogues appear comparable.

In this study, patients eligible and consented for ESG will be retrospectively matched against a group of patients who were previously placed on GLP-1 analogue treatment for class 1 and 2 obesity.

The primary outcome of the study will be total body weight loss at 1-year. We will also examine the short-term weight loss outcomes, metabolic outcomes, as well as healthcare costs between the 2 groups. Our hypothesis is that ESG will be non-inferior to GLP-1 analogues in weight loss and metabolic outcomes, with reduced healthcare costs, given the avoidance of repeated dosing.

ELIGIBILITY:
Inclusion Criteria:

* Patients with classes 1 (BMI 27.5 to 34.9) and 2 (BMI 35 to 39.9) obesity in accordance with the World Health Organisation recommendations but modified to the interventional thresholds recommended for Asian populations

Exclusion Criteria:

* Patients with class 3 obesity and above (BMI > 40.0)
* Patients with contraindications to GLP-1 analogues
* Patients with contraindications to endoscopic sleeve gastroplasty
* Patients with previous bariatric or upper gastrointestinal surgery

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-10-07 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Total body weight loss | 1-year
  Percentage total body weight loss

SECONDARY OUTCOMES:
Short-term weight loss | 3-months
  Percentage total body weight loss
Short-term weight loss | 6-months
  Percentage total body weight loss
Short-term weight loss | 9-months
  Percentage total body weight loss
Healthcare costs | 1-year
  Patient costs associated with procedure, hospital stay, outpatient visits and pharmacological treatment
Metabolic outcomes | 3-months, 6-months, 9-months, 12-months
  HbA1c values

CONTACTS AND LOCATIONS:
Locations (1):
- Sengkang General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No